CLINICAL TRIAL: NCT00204087
Title: Psychological Intervention for Persons at Risk of Psychosis in the Early Initial Prodromal State
Brief Title: Psychological Intervention for Persons in the Early Initial Prodromal State
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cologne (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); German Research Network On Schizophrenia (Network); Department of Psychiatry University of Bonn (Other); Heinrich-Heine University, Duesseldorf (Other); Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01 GI 9935 - P 1.1.2
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-01-12 (Estimated); Status verified 1999-06

CONDITIONS: Schizophrenia; Psychosis
Keywords: Schizophrenia; Psychosis; Prodrome; Early Initial Prodromal State; Early Intervention; Cognitive Behavioral Therapy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT)
Behavioral: Supportive Counselling (SC)

SUMMARY:
The purpose of this randomized controlled trial is to develop a cognitive behavioral therapy (CBT) for persons with at risk mental states in the early initial prodromal state and to evaluate CBT in comparison to supportive counselling (SC).It is hypothesized that CBT is more effective than SC on transition to subthreshold psychosis, psychosis and schizophrenia as well as on prodromal symptoms and social adjustment.

DETAILED DESCRIPTION:
Several studies indicated that self-perceived cognitive thought and perception deficits (basic symptoms), negative symptoms, anxiety, depressive symptoms and social stagnation or social decline are usually present years before the first episode of schizophrenia appears. It is also known that delayed treatment of schizophrenia correlates with a poor prognosis, low compliance and high family burden. As consequence of these findings, for the first time we developed a cognitive behavioral therapy (CBT) for persons at risk for psychosis in the early initial prodromal state. The early initial prodromal state was defined by the presence of self-perseived neuropsychological deficits, which were found to be predictive for transition to psychosis and by the presence of clinical relevant decline of functioning in combination with that of clinical management (CM). Is CBT more effective than CM with regard to the three aims of intervention 1. transition to psychosis, 2. improvement of prodromal symptoms, 3. prevention of social decline/stagnation, ? A randomized controlled trail is used to compare the efficacy of CBT with that of supportive counselling (SC). Patients are randomized to receive either CBT or SC over a 12 months period. CBT comprises of individual and group therapy as well as cognitive remediation and psychoeducation for key persons. SC should provide regular supportive contacts for the patient. No CBT strategies are allowed to be systematically applied in SC.

ELIGIBILITY:
Inclusion Criteria:

1. General criteria

   * Age between 17 and 36 years
   * male or female, in- or outpatients
   * written informed consent, for patients below 18 years also signed by their parents
2. Special criteria (presented within the last three months prior to the study)

   1. Self-experienced neuropsychological deficits (basic symptoms)

      * Thought interferences
      * Compulsory like perseverance of thoughts
      * Thought pressure
      * Thought blockages
      * Disturbances of receptive language, either heard or read
      * Decreased ability to discriminate between ideas and perception, fantasy and true memories
      * Unstable ideas of reference (subject-centrism)
      * Derealisation
      * Visual perceptual disturbances (blurred vision, transitory blindness, partial seeing, hypersensitivity of light, etc..)
      * Acoustic perceptual disturbances (hypersensitivity to sounds or noise (hypersensitivity to sounds or noise, acoasms, etc.) AND/OR
   2. Reduction in the Global Assessment of Functioning Score (DSM IV) of at least 30 points (within the past year) and at least one of the following risk factors:

      * First-degree relative with a lifetime-diagnosis of schizophrenia or
      * a schizophrenia spectrum disorder
      * Pre-or perinatal complications

Exclusion Criteria:

* Attenuated or transient positive symptomes
* Present or past diagnosis of a schizophrenic, schizophreniform, schizoaffective, delusional or bipolar according to DSM IV
* Present or past diagnosis a brief psychotic disorder according to DSM IV with a duration of more than one week or within the last 4 weeks regardless of its duration
* Diagnosis of delirium, dementia, amnestic or other cognitive disorder, mental retardation psychiatric disorder due to a somatic factor or related to the consumption of psychotropic substances according DSM IV
* Alcohol- or drug abuse within the last three months prior to inclusion according to DSM IV
* Deases of the central nervous system (inflammatory, traumatic, epilepsy etc.)

Ages: 17 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126
Dates: Start 2001-01; Study Completion 2005-06

PRIMARY OUTCOMES:
transition to subthreshold psychosis (and psychosis or schizophrenia)

SECONDARY OUTCOMES:
improvement of prodromal symptoms (basic symptoms, depression, anxiety)
social adjustment

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bechdolf, Dr., Study Chair — Department of Psychiatry and Psychotherapy, University of Cologne
Locations (1):
- Department of Psychiatry and Psychotherapy, University of Cologne, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Wessels H, Wagner M, Kuhr K, Berning J, Putzfeld V, Janssen B, Bottlender R, Maurer K, Moller HJ, Gaebel W, Hafner H, Maier W, Klosterkotter J, Bechdolf A. Predictors of treatment response to psychological interventions in people at clinical high risk of first-episode psychosis. Early Interv Psychiatry. 2019 Feb;13(1):120-127. doi: 10.1111/eip.12460. Epub 2017 Jul 4. PMID 28675695
- [Derived] Bechdolf A, Wagner M, Ruhrmann S, Harrigan S, Putzfeld V, Pukrop R, Brockhaus-Dumke A, Berning J, Janssen B, Decker P, Bottlender R, Maurer K, Moller HJ, Gaebel W, Hafner H, Maier W, Klosterkotter J. Preventing progression to first-episode psychosis in early initial prodromal states. Br J Psychiatry. 2012 Jan;200(1):22-9. doi: 10.1192/bjp.bp.109.066357. Epub 2011 Nov 10. PMID 22075649
- See also: Click here for more information about this study: Psychological intervention for persons at risk of psychosis in the early initial prodromal state — http://www.kompetenznetz-schizophrenie.de
- See also: Related Info — http://www.fetz.de